CLINICAL TRIAL: NCT01814657
Title: Optimizing Patient Analgesic Experience During IVF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 00029750
Record Dates: First submitted 2013-03-08; First posted 2013-03-20 (Estimated); Last update posted 2022-07-18 (Actual); Status verified 2014-12

CONDITIONS: Infertility
Keywords: Infertility
MeSH Terms: conditions — Infertility | interventions — Lidocaine; Solutions

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Normal Saline (Placebo Comparator): Conscious sedation and sterile normal saline (placebo) paracervical block
  Interventions: Drug: Sterile Normal Saline%
- Lidocaine (Active Comparator): Conscious sedation and Lidocaine hydrochloride 1% solution paracervical block
  Interventions: Drug: Lidocaine hydrochloride (HCl) 1% solution

INTERVENTIONS:
Drug: Lidocaine hydrochloride (HCl) 1% solution — Comparison of paracervical block using Lidocaine versus Normal Saline placebo in patients undergoing oocyte retrieval during IVF.
  Other Names: Xylocaine
  Arms: Lidocaine
Drug: Sterile Normal Saline% — Sterile normal saline used as placebo for lidocaine hydrochloride (HCl)1% solution
  Other Names: Sterile Normal Saline
  Arms: Normal Saline

SUMMARY:
This study is for patients undergoing In Vitro Fertilization (IVF). The investigators are studying the best way to control pain during the egg retrieval process. The egg retrieval involves passing a needle under ultrasound guidance through the vagina into the ovaries to remove eggs that are to be later fertilized. Patients often report this as very uncomfortable.

Different fertility clinics across the country use different methods of pain control. All clinics will use intravenous medication to control pain, while some may or may not use local anaesthetic (freezing) in the vagina. Our goal is to find the best way to control pain. Since local anaesthetic injection involves multiple needle punctures and may be painful, the investigators are unsure if local anaesthetic is necessary in addition to the intravenous pain medication.

The investigators will conduct a randomized trial where all patients will receive intravenous pain medication, but some will receive local anaesthetic injection and some will receive placebo injection. Patients will be asked to complete a questionnaire on their pain experience after oocyte retrieval. The investigators will then analyze the data and determine whether local anaesthetic actually improves pain when patients are already receiving intravenous pain medications. Through our study, the investigators aim to improve the pain experience of all women undergoing IVF in the future.

DETAILED DESCRIPTION:
Background:

A UK telephone survey (Bokhari, 1999) showed that during TUGOR, 48% of UK fertility centers were using conscious sedation, 29% general anaesthesia, 12% conscious sedation with regional anaesthesia (neuraxial block or PCB), and 2% regional anaesthesia alone. A review article (Blahos 2009) details the many different types of anaesthesia used during TUGOR. These may include combinations of the following: general anaesthesia, regional anaesthesia, local anaesthesia, conscious sedation, and alternative methods of anaesthesia (electro-acupuncture, patient controlled sedation). No recent studies were found detailing the frequency of each of the various anaesthetic options in use at fertility centers across North American.

A prospective, randomized, double-blind and placebo controlled study (Ng, 1999) showed that paracervical block combined with conscious sedation was superior to conscious sedation alone. This study used a combination of drugs (mepiridine and diazepam) not used at our center. The use of fentanyl and midazolam was first described by Harrison in 1992 for conscious sedation. In 2001 Sephton et al published a cross over audit of patient preferences comparing mepiridine, diazepam and promethazine to fentanyl and midazolam, showing superiority of fentanyl and midazolam. Midazolam has sedative and amnestic properties, whereas diazepam has no amnestic properties. The amnestic properties of midazolam make it a superior medication for overall patient experience during TUGOR, as they are less likely to recall potentially painful parts of their procedure. Midazolam has also been shown to act synergistically with fentanyl, thereby decreasing not only the actual pain recalled, but the actual pain experienced by patients. Since the only randomized control trial demonstrating the benefits of paracervical block was performed using mepiridine and diazepam, we intend to repeat the study using the superior combination of fentanyl and midazolam.

Study Rationale:

The oocyte retrieval may be the most painful part of fertility treatment. Our goal is to minimize patient discomfort and improve overall patient experience during fertility treatments. We do not know if PCB improves pain scores in the era of wider use of fentanyl and midazolam for sedation. Fertility centres may be subjecting their patients to a painful PCB injection without proven benefit. This study aims to assess whether a PCB in addition to conscious sedation can be abandoned without impacting the patient's overall pain experience.

Study Objective:

The objective is to compare whether conscious sedation alone is as effective as paracervical block plus conscious sedation in controlling pain during oocyte retrieval

Study Question:

Is conscious sedation alone as effective as paracervical block plus conscious sedation in controlling pain during oocyte retrieval?

Overview of the Trial Design This study is designed to be a placebo-controlled, randomised, double blind trial to compare whether conscious sedation with a normal saline paracervical block (placebo) is as effective as conscious sedation with a lidocaine paracervical block in controlling pain during oocyte retrieval. A total of 300 women will randomly be assigned in a 1:1 ratio, after consenting to study participation. Short-Form McGill Pain scores will be assessed in study subjects.

Study Population:

Women presenting for oocyte retrieval after a cycle of IVF stimulation at the University of Alberta Regional Fertility Centre

Study Design:

Women consenting to participate in the study will be randomly allocated to one of two groups. The control group will receive conscious sedation with a placebo (normal saline) paracervical block (PCB). The study group will receive conscious sedation with a local anaesthetic (lidocaine 1%) PCB. Computer generated randomisation will be used to determine group allocation. Group allocation will be concealed using opaque envelopes to ensure blinding. An OR nurse will prepare the PCB syringe with either lidocaine or normal saline depending on the patient's allocation. The contents of the PCB will remain blinded from the physician performing the TUGOR and the patient.

The fertility centre's routine for TUGOR is as follows: Initially conscious sedation is administered by OR nursing staff according to the patient's weight (midazolam 1 - 2 mg and fentanyl 50 - 75 ug IV). This is followed by the PCB 5 minutes later. Additional fentanyl is administered throughout the procedure as required to ensure patient comfort. The oocyte retrieval proceeds once the PCB is completed. Following the oocyte retrieval and when the conscious sedation has worn off; the patient will be assessed before discharge. Once the discharge criteria have been met, the validated and standardized Short-Form McGill Pain Questionnaire will be used to objectively measure the pain experienced during the TUGOR. All study participants will be required to rate the pain experience during the procedure. The attending nurse is required to record all adverse events from the procedure as part of her clinical duties. Embryology information, i.e. fertilization, embryo grading, development and frozen rates will be recorded to assess whether PCB affects this aspect of ART. Additional information will be obtained by reviewing participants' clinic charts nine months post-procedure to determine secondary outcomes, i.e. live birth rates. Animal mouse models in the past have shown local anaesthetic to adversely affect fertilization and embryo development (Schnell, 1992). No adverse effects on human embryos from lidocaine have ever been demonstrated (Wikland 1990), however assessing embryo quality and birth outcomes has been the standard when conducting studies assessing the use of PCB

Setting:

Academic referral fertility centre

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing oocyte retrieval who have consented to participation
* Only the first ART cycle will be included

Exclusion Criteria:

* History of drug sensitivity to local anaesthetic agents
* Women with any chronic pain syndrome

Ages: 21 Years to 43 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 308 (Actual)
Dates: Start 2013-03; Primary Completion 2015-11-07 (Actual); Study Completion 2015-11-07 (Actual)

PRIMARY OUTCOMES:
Pain scores rated on SF-MPQ | Data collection is scheduled to proceed until 308 participants have been recruited which is anticipated to take up to 2 years.
  Score rating will be done before the patient is discharged following oocyte retrieval.

SECONDARY OUTCOMES:
Embryology data | Assessed within 7 days of oocyte retrieval
  Recorded as number of embryos obtained. Number of embryos transferred. The decision to transfer Day 3 embryos or Day 5 blastocysts. Number of embryos or blastocysts frozen. Embryological grading of all embryos or blastocysts either transferred or frozen.

OTHER OUTCOMES:
Live Birth Rates | Within 12 months of oocyte retrieval
  Recorded as the number of infants born alive to the patient that resulted from embryos transferred during this study.

CONTACTS AND LOCATIONS:
Overall Officials: Tarek Motan, MB ChB, Principal Investigator — University of Alberta
Locations (1):
- Fertility and Womens Endocrine Clinic, Edmonton, Alberta, Canada

REFERENCES:
- [Background] Ng EH, Tang OS, Chui DK, Ho PC. A prospective, randomized, double-blind and placebo-controlled study to assess the efficacy of paracervical block in the pain relief during egg collection in IVF. Hum Reprod. 1999 Nov;14(11):2783-7. doi: 10.1093/humrep/14.11.2783. PMID 10548622
- [Background] Bhattacharya S, MacLennan F, Hamilton MP, Templeton A. How effective is patient-controlled analgesia? A randomized comparison of two protocols for pain relief during oocyte recovery. Hum Reprod. 1997 Jul;12(7):1440-2. doi: 10.1093/humrep/12.7.1440. PMID 9262274
- [Background] Elkington NM, Kehoe J, Acharya U. Intravenous sedation in assisted conception units: a UK survey. Hum Fertil (Camb). 2003 May;6(2):74-6. doi: 10.1080/1464770312331369083. PMID 12869788
- [Background] Bokhari A, Pollard BJ. Anaesthesia for assisted conception: a survey of UK practice. Eur J Anaesthesiol. 1999 Apr;16(4):225-30. doi: 10.1046/j.1365-2346.1999.00461.x. PMID 10234491
- [Background] Vlahos NF, Giannakikou I, Vlachos A, Vitoratos N. Analgesia and anesthesia for assisted reproductive technologies. Int J Gynaecol Obstet. 2009 Jun;105(3):201-5. doi: 10.1016/j.ijgo.2009.01.017. Epub 2009 Feb 26. PMID 19249049
- [Background] Sephton VC, Shaw A, Cowan CM, Thomas K, Wood S, Barclay PM, Kingsland CR. Sedation and analgesia for transvaginal oocyte retrieval: an audit resulting in a change of clinical practice. Hum Fertil (Camb). 2001;4(2):94-8. doi: 10.1080/1464727012000199361. PMID 11591263
- [Background] Harrison RF, Barry-Kinsella C, Drudy L, Gordon A, Hannon K, Hennelly B, Keogh I, Kondaveeti U, Nargund G, Verso J. An Irish out-patient based in-vitro fertilisation service. Ir Med J. 1992 Jun;85(2):63-5. PMID 1628945
- [Background] Gohar J, Lunenfeld E, Potashnik G, Glezerman M. The use of sedation only during oocyte retrieval for in vitro fertilization: patients' pain self-assessments versus doctors' evaluations. J Assist Reprod Genet. 1993 Oct;10(7):476-8. doi: 10.1007/BF01212936. No abstract available. PMID 8069089
- [Background] Wikland M, Evers H, Jakobsson AH, Sandqvist U, Sjoblom P. The concentration of lidocaine in follicular fluid when used for paracervical block in a human IVF-ET programme. Hum Reprod. 1990 Nov;5(8):920-3. doi: 10.1093/oxfordjournals.humrep.a137220. PMID 2081803
- [Background] Schnell VL, Sacco AG, Savoy-Moore RT, Ataya KM, Moghissi KS. Effects of oocyte exposure to local anesthetics on in vitro fertilization and embryo development in the mouse. Reprod Toxicol. 1992;6(4):323-7. doi: 10.1016/0890-6238(92)90195-y. PMID 1521005